CLINICAL TRIAL: NCT00708578
Title: Insulin Glargine Combined With Sulfonylurea Versus Metformin in Patients With Type 2 Diabetes: A Randomized, Controlled Trial.
Brief Title: Optimal Oral Hypoglycaemic Agents (OHA) for Combination With Insulin Glargine (Sulfonylurea vs. Metformin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_02670
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Administration of 4 mg of Glimepiride with Insulin Glargine
  Interventions: Drug: Glimepiride; Drug: Insulin Glargine
- 2 (Active Comparator): Administration of 1500 mg of Metformin with Insulin Glargine
  Interventions: Drug: Metformin; Drug: Insulin Glargine
- 3 (Experimental): Administration of a combination of 4mg Glimepiride plus 1000mg Metformin with Insulin Glargine
  Interventions: Drug: Glimepiride; Drug: Metformin; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Glimepiride — Once a day before breakfast
  Arms: 1; 3
Drug: Metformin — After breakfast and supper
  Arms: 2; 3
Drug: Insulin Glargine — Injection in the morning

SUMMARY:
Primary objective:

To find out an optimal regimen of OHA (oral hypoglycaemic agents) in combination with insulin glargine (metformin, glimepiride or metformin+glimepiride) by measuring HbA1c level

Secondary objective:

To compare the incidence of hypoglycemia in each treatment group

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 6 months
* Treated with maximal, tolerable dose of metformin (≥ 1000mg/day) and sulfonylurea (glimepiride≥ 4 mg/day or equivalent dose of other SU) for at least 3 months prior to the screening visit
* 7.0 < HbA1c < 11 %
* Fasting serum C-peptide > 0.33 nmol/L
* BMI < 30 kg/m²
* Patients who is willing to monitor BG using SMBG

Exclusion Criteria:

* Type 1 Diabetes
* Clinical evidence of active liver disease, or serum ALT 3 times the upper limit of the normal range
* Serum creatinine: ≥ 1.5 mg/dl for males, ≥ 1.4 mg/dl for females
* Active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before study entry or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study (an optic fundus examination should have been performed in the 2 years prior to study entry)
* History of alcohol or other substance abuse
* Pregnancy or not using contraceptive in childbearing aged women
* Breast feeding women
* History of hypersensitivity to the study drugs or to drugs with a similar chemical structure
* Treatment with any medication including corticosteroid or herbal medicines that can affect blood glucose level within 3 months prior to study entry except metformin and sulfonylurea.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HbA1c values | At baseline to end of treatment

SECONDARY OUTCOMES:
Hypoglycemia events | From inclusion to end of study
Percentage of patients with HbA1c < 7% | At the end of the study
Fasting Blood Glucose level | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Ahn, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Seoul, South Korea

REFERENCES:
- [Derived] Park CY, Kang JG, Chon S, Noh J, Oh SJ, Lee CB, Park SW. Comparison between the therapeutic effect of metformin, glimepiride and their combination as an add-on treatment to insulin glargine in uncontrolled patients with type 2 diabetes. PLoS One. 2014 Mar 10;9(3):e87799. doi: 10.1371/journal.pone.0087799. eCollection 2014. PMID 24614911